CLINICAL TRIAL: NCT06531629
Title: Risk-based Screen and Prognostic Analysis for Second Primary Malignancies in Kidney Cancer Patients: A Retrospective Cohort Study Based on Large-scale Population and Mendelian Randomization Analysis
Brief Title: Risk-based Screen and Prognostic Analysis for Second Primary Malignancies in Kidney Cancer Patients
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, GONG Kan, Chief physician, Peking University First Hospital
Other Study IDs: 2024#07-03
Record Dates: First submitted 2024-07-27; First posted 2024-08-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Kidney Cancer
Keywords: Kidney cancer; Prediction model; Prognosis; Risk factors; Second primary malignancy
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms, Second Primary | interventions — Surgical Procedures, Operative; Radiotherapy; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney cancer patients with second primary malignancy (SPM): Patients diagnosed with first primary kidney cancer and second primary malignancy between 2000 and 2020
  Interventions: Procedure: Surgery, radiation therapy and chemotherapy
- Kidney cancer patients without SPM: Patients diagnosed with only first primary kidney cancer between 2000 and 2020
  Interventions: Procedure: Surgery, radiation therapy and chemotherapy

INTERVENTIONS:
Procedure: Surgery, radiation therapy and chemotherapy — Surgery, radiation therapy and chemotherapy

SUMMARY:
Second primary malignancy (SPM) significantly impacts the survival and prognosis of patients. This study endeavors to identify risk and prognostic factors associated with SPM after first primary kidney cancer and construct predictive nomograms.

DETAILED DESCRIPTION:
In recent years, with the advancement of cancer treatment techniques and the prolonged survival of patients, the prevalence of Second primary malignancy (SPM) has been escalating, emerging as a significant health issue among cancer survivors. The goal of this study is to identify risk and prognostic factors associated with SPM after first primary kidney cancer and construct nomograms to provide clinical evidence. The main questions this study aims to answer are: (1) What are the risk factors associated with the prevalence of SPM after kidney cancer? (2) What are the prognostic factors associated with the overall survival (OS) of kidney cancer patients with SPM? (3) How to accurately predict the probability of developing SPM after kidney cancer and the OS of kidney cancer patients with SPM? In this retrospective population-based cohort study, Patients diagnosed with first primary kidney cancer between 2000 and 2020 were retrospectively enrolled from the Surveillance, Epidemiology, and End Results (SEER) database. Researchers will concentrate on the risk and prognostic factors of SPM after kidney cancer, and develop nomograms to forecast the development and overall survival (OS) of SPM after kidney cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Diagnosed age was between 18 and 80 years old
* (2) Diagnosed histologically confirmed as first primary kidney cancer
* (3) The staging of kidney cancer was early or localized advanced (T1/2/3N0M0)
* (4) Detailed survival data and follow-up information should be provided

Exclusion Criteria:

* (1) Histological conformation for diagnosis was unavailable
* (2) The type of reporting source was "Death certificate only" or "Autopsy only"
* (3) Patients with other malignancies before the diagnosis of primary kidney cancer
* (4) The staging of kidney cancer was not early or localized advanced (T1/2/3N0M0)
* (5) Diagnosis interval between first primary malignancy (FPM) and second primary malignancy (SPM) was less than 6 months
* (6) The information was not complete

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospectively reviewing data were obtained from the Surveillance, Epidemiology, and End Results (SEER) database (https://seer.cancer.gov/) from 2000-2020 using SEER Stat 8.4.1. This study was based on the Surveillance, Epidemiology, and End Results (SEER) database, which contains the population-based data from 17 Registries covering approximately 26.5% of the U.S. population.The eligible kidney cancer patients were identified from the SEER database.
Sampling Method: Non-Probability Sample
Enrollment: 72408 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Developing a second primary malignancy (SPM) | This time was calculated as the time interval from the diagnosis of first primary kidney cancer to the diagnosis of second primary malignancy, assessed up to 20 years.
  This time was calculated as the time interval from the diagnosis of first primary kidney cancer to the diagnosis of second primary malignancy.
Overall survival (OS) | From the date of diagnosis of the second primary malignancy to the date of death from any cause or the data of last follow-up, whichever came first, assessed up to 20 years.
  OS was calculated as the time interval from the diagnosis of the second primary malignancy to death or the time to the last follow-up.

SECONDARY OUTCOMES:
Cancer-specific survival (CSS) | From date of diagnosis of the second primary malignancy until the date of death from the same disease or the date of last follow-up, whichever came first, assessed up to 20 years.
  CSS was calculated as the time interval from the diagnosis of the second primary malignancy to death from the same disease or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Gong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China